CLINICAL TRIAL: NCT04050514
Title: Side Effects of Two Different Mandibular Advancement Devices (MAD) in the Treatment of Snoring and Obstructive Sleep Apnea Syndrome (OSAS)
Brief Title: Side Effects of Mandibular Advancement Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 001072019
Record Dates: First submitted 2019-08-01; First posted 2019-08-08 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Obstructive Sleep Apnea Syndrome; Temporomandibular Disorders
Keywords: side effects; mandibular advancement device; clinical intervention; snoring; treatment
MeSH Terms: conditions — Sleep Apnea, Obstructive; Temporomandibular Joint Disorders; Snoring

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized two-arm study with active control group, stratified by gender.
Who Masked: Participant, Outcomes Assessor
Masking Description: Unblinded with respect to the examiner, blinded to the patient and statisticians in the evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H-MAD, hinge system according to Herbst (Experimental): Patients with snoring and OSAS. Therapy with MAD type H-MAD with lateral hinges according to Herbst.
  Bite elevation 2 mm interocclusal distance with a lower jaw advancement of 5 mm
  Interventions: Device: H-MAD with a hinge system according to Herbst
- F-MAD, SomnoDent Fusion (Active Comparator): Patients with snoring and OSAS,Fusion MAD with sliding side wings (F-MAD). Bite elevation 5 mm interocclusal distance with a lower jaw advancement of 5 mm
  Interventions: Device: H-MAD with a hinge system according to Herbst

INTERVENTIONS:
Device: H-MAD with a hinge system according to Herbst — The randomized grouping into blocks at a ratio of 1: 1 takes place over sealed envelopes containing the allocation key for the respective MAD. The assignment is stratified according to gender because gender is a strong predictor of sleep disorders and also temporomandibular dysfunctions Integration of the MAD (start of treatment) The laboratory-made MAD (F-MAD / H-MAD) is integrated and checked for a comfortable fit. The patient is instructed to always wear the splint during sleep.
  All patients receive an extended guide to jaw gymnastics with the instruction to do it in the morning after waking up and in the evening before falling asleep.
  Four weeks after incorporation, the titration phase begins, the slow adjustment of mandibular advancement to optimize sleep medical parameters while minimizing unwanted side effects.
  Control appointments take place after four weeks, six months, one year and two years after insertion of the MAD

SUMMARY:
Sleep-related breathing disorders (SBAS) are one of the most common causes of non-restorative sleep.

Sleep therapy options include positive pressure ventilation with continuous positive airway pressure (CPAP) masks, mandibular advancement of the mandible with mandibular advancement devices (MAD), back restraining, weight reduction, ear, nose and throat surgical procedures, bimaxillary or mandibular remodeling osteotomies, and neurostimulation procedures N. hypoglossal. In mild to moderate obstructive sleep apnea syndrome (OSAS), MAD, back suppression and weight reduction are potential treatment options. This study aims to identify possible side effects in the temporomandibular system that occur during nocturnal support of a mandibular arch over two years. Two different MADs are compared in terms of construction, height (bite elevation) and protrusion mechanics: the H-MAD with an hinge system according to Herbst and the SomnoDent Fusion ™ MAD (called F-MAD) with sliding side wings.

In addition, it is to be evaluated whether hinge system according to Herbst as a protrusion-controlling element and the reduction of the splint body for a reduced bite elevation leads to a significant reduction of side effects compared to the F-MAD.

DETAILED DESCRIPTION:
Sleep-related breathing disorders (SBAS), particularly obstructive sleep apnea syndrome (OSAS), are one of the most common causes of non-restorative sleep. Disturbances of sleep disorders include apneas and hypopneas associated with either or not pharyngeal obstruction and hypoventilation. Depending on the type of respiratory disorder present, they are associated with hypoxemia and may cause hypercapnia or acidosis The consequences of obstructive narrowing of the pharynx are far-reaching. Studies have shown that patients with OSAS have comorbidities such as neurological complaints, heart attacks, dementia, cardiovascular complaints, myocardial infarction, and a higher mortality rate.

Sleep fragmentation caused by respiratory disorders during sleep and wakefulness reactions (arousals) can lead to daytime sleepiness and concentration disorders. In the longer term untreated arousals and apneas are associated with an increased risk for arterial hypertension, stroke, myocardial infarction, diabetes mellitus and libido loss.

OSAS management includes positive pressure ventilation with continuous positive airway pressure (CPAP) masks, mandibular advancement of the mandible with mandibular advancement devices (MAD), weight loss, ear, nose and throat surgical procedures, bimaxillary or mandibular remodeling osteotomies, and neurostimulation procedures of the hypoglossal nerve.

Several studies have shown that the use of MADs is inferior in reducing the severity of OSAS in comparison to CPAP therapy, but its efficacy is comparable and preferred by patients in mild to moderate OSAS.

Due to the forward displacement of the lower jaw for several hours at night, similar symptoms as in temporomandibular dysfunction (TMD) patients may occur. The symptoms may be pain or stiffness on the masticatory muscles or temporomandibular joints.

This study aims to identify possible side effects in the temporomandibular system that occur during the course of two years of nocturnal MAD delivery. Two different appliance systems are compared in terms of construction height (bite elevation) and protrusion mechanics: the H-MAD ™ with a hinge system according to Herbst and the SomnoDent Fusion ™ (called F-MAD) with sliding side wings.

ELIGIBILITY:
Inclusion Criteria:

* Patients with medical indication for mandibular protrusion (MAD) due to OSAS
* therapy request for snoring
* Body Mass Index (BMI) ≤ 35
* mandibular protrusion of 5 mm possible
* at least 8 remaining teeth or 4 implants per jaw
* fixed dentures and stable
* removable partial denture, at least support up to the area of the 2nd premolars on both sides
* business ability and the existence of the signed declaration of consent

Exclusion Criteria:

* polyarthritis
* fibromyalgia, neuralgia
* central sleep apnea syndrome
* untreated generalized periodontitis
* chronic dysfunctional pain degree 3-4
* long-term use of psychotropics and analgesics (> 4 weeks)
* pregnancy
* participation in another interventional clinical study (currently up to three months before inclusion)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
change orofacial pain: numeric rating scale (NRS; 0-10) | 4 weeks, six months, one year, two years
  change of orofacial pain after applying the MAD measured by numeric rating scale (NRS; 0-10, 0: no pain, 10: worst imaginable pain)

SECONDARY OUTCOMES:
pressure pain points on palpation | 4 weeks, six months, one year, two years
  number of pressure pain points on palpation of the masticatory muscles and in the area of the temporomandibular joints according to the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD)
number of posterior contact points | 4 weeks, six months, one year, two years
  change of the number of occluding posterior teeth

OTHER OUTCOMES:
change in sleep quality: Pittsburgh Sleep Quality Index (PSQI, 0-21, < 5: good sleep) | 4 weeks, six months, one year, two years
  change in sleep quality after applying the MAD measured by Pittsburgh Sleep Quality Index retrospectively asks for a four-week period the incidence of sleep disturbing events, sleep quality assessment, sleep habits, sleep latency and sleep duration, sleeping medication use.
change in daytime sleepiness: Epworth Sleepiness Scale (ESS, 0-24, <11 no daytime sleepiness) | 4 weeks, six months, one year, two years
  Change in daytime sleepiness measured by Epworth Sleepiness Scale. ESS is a short questionnaire for the detection of daytime sleepiness. (ESS, 0-24, <11 no daytime sleepiness)
change in oral health-related quality of life: Oral Health Impact profile (OHIP-5) (0-20) | 4 weeks, six months, one year, two years
  Oral Health Impact profile (OHIP-5) is a measurement tool for assessing the oral health-related quality of life in adults. It consists of 5 questions for functional limitation, physical pain, psychological discomfort, physical disability, social disability
change in chronic pain: Graded Chronic Pain Scale (GCPS) questionnaire (0-4) | 4 weeks, six months, one year, two years
  Graded Chronic Pain Scale (GCPS) questionnaire records pain intensity and the presence of functional or dysfunctional chronic pain. Three subscale scores (characteristic pain intensity, disability score, and the disability points score) are used to classify subjects into 1 of the 5 pain severity grades: grade 0 for no pain, grade 1displays low disability, low intensity, grade 2 displays low disability but high intensity, grade 3 displays high disability,moderately limiting and grade 4 displays high disability and severely limiting.

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Bernhardt, Prof., Principal Investigator — University Medicine Greifswald
Locations (9):
- Germany (9):
  - Dental Office Dr. Krumholz, Frankfurt
  - Dental Office Dr. Schlieper, Hamburg
  - Dental Office Dr. Hauschild, Isernhagen-Süd
  - Zahnarztpraxis Weststadt, Karlsruhe
  - Dental Office Dr. Kares, Saarbrücken
  - Dental Office Dr. Heckmann, Saarlouis
  - Dental Office Dr. Meyer, Solingen
  - Dental Office Dr. Nauert, Sulzbach
  - Mund-Zahn-Kiefer-Klinik, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Haviv Y, Rettman A, Aframian D, Sharav Y, Benoliel R. Myofascial pain: an open study on the pharmacotherapeutic response to stepped treatment with tricyclic antidepressants and gabapentin. J Oral Facial Pain Headache. 2015 Spring;29(2):144-51. doi: 10.11607/ofph.1408. PMID 25905532
- [Background] Ringqvist M, Walker-Engstrom ML, Tegelberg A, Ringqvist I. Dental and skeletal changes after 4 years of obstructive sleep apnea treatment with a mandibular advancement device: a prospective, randomized study. Am J Orthod Dentofacial Orthop. 2003 Jul;124(1):53-60. doi: 10.1016/s0889-5406(03)00240-3. PMID 12867898
- [Background] Perez CV, de Leeuw R, Okeson JP, Carlson CR, Li HF, Bush HM, Falace DA. The incidence and prevalence of temporomandibular disorders and posterior open bite in patients receiving mandibular advancement device therapy for obstructive sleep apnea. Sleep Breath. 2013 Mar;17(1):323-32. doi: 10.1007/s11325-012-0695-1. Epub 2012 Apr 4. PMID 22477031
- [Background] Gesch D, Bernhardt O, Kocher T, John U, Hensel E, Alte D. Association of malocclusion and functional occlusion with signs of temporomandibular disorders in adults: results of the population-based study of health in Pomerania. Angle Orthod. 2004 Aug;74(4):512-20. doi: 10.1043/0003-3219(2004)0742.0.CO;2. PMID 15387030
- [Background] Doff MH, Hoekema A, Pruim GJ, Huddleston Slater JJ, Stegenga B. Long-term oral-appliance therapy in obstructive sleep apnea: a cephalometric study of craniofacial changes. J Dent. 2010 Dec;38(12):1010-8. doi: 10.1016/j.jdent.2010.08.018. Epub 2010 Sep 8. PMID 20831889
- [Background] Bacon W, Tschill P, Sforza E, Krieger J. [A device for mandibular advancement in respiratory disorders of sleep. Clinical study]. Orthod Fr. 2000 Dec;71(4):295-302. French. PMID 11196228
- [Derived] Bernhardt O, Giannakopoulos NN, Kares H, Meyer A, Nurnberger CM, Ruge S, Schwahn C, Schlieper J, Yousif S, Zenner H, Kanzow P. Side effects of mandibular advancement devices in obstructive sleep apnea patients - observational results of a randomized controlled trial. Sleep Breath. 2026 Feb 3;30(1):32. doi: 10.1007/s11325-026-03576-4. PMID 41634250

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT04050514/Prot_SAP_000.pdf